CLINICAL TRIAL: NCT05268185
Title: A Randomized Controlled Trial to Assess Differences Between Mixing or Matching of Moderna and Pfizer Booster Vaccines for Covid-19 Citizen Science (CCS) Participants
Brief Title: The BOOSTED (Booster Options Or Switching Tested for Effectiveness and Downsides Study) Trial (COVID-19)
Acronym: BOOSTED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-35575
Record Dates: First submitted 2022-02-28; First posted 2022-03-07 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Vaccine Reaction; COVID-19 Pandemic
Keywords: COVID-19; Remote; Vaccine; COVID-19 Citizen Science Study
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Moderna Booster Recommendation (Active Comparator): Participants assigned to this arm will be recommended to receive the Moderna vaccine for their Covid-19 booster shot.
  Interventions: Behavioral: Moderna Booster Vaccine
- Pfizer Booster Recommendation (Active Comparator): Participants assigned to this arm will be recommended to receive the Pfizer vaccine for their Covid-19 booster shot.
  Interventions: Behavioral: Pfizer Booster Vaccine

INTERVENTIONS:
Behavioral: Moderna Booster Vaccine — Participants assigned to this intervention will be given the recommendation to receive the Moderna vaccine for their Covid-19 booster shot. The study team will not be administering vaccines to the participants; participants must have equal access to both the Pfizer and Moderna booster vaccines to be eligible for this study. According to current FDA recommendations, Moderna booster (0.25 mL) may be administered as a heterologous booster dose following completion of primary vaccination with another authorized or approved COVID-19 vaccine. The dosing interval for the heterologous booster dose is the same as that authorized for a booster dose of the vaccine used for primary vaccination.
  Arms: Moderna Booster Recommendation
Behavioral: Pfizer Booster Vaccine — Participants assigned to this intervention will be given the recommendation to receive the Pfizer vaccine for their Covid-19 booster shot. The study team will not be administering vaccines to the participants; participants must have equal access to both the Pfizer and Moderna booster vaccines to be eligible for this study. According to current FDA recommendations, the Pfizer booster (0.30 mL) may be administered as a heterologous booster dose following completion of primary vaccination with another authorized or approved COVID-19 vaccine. The dosing interval for the heterologous booster dose is the same as that authorized for a booster dose of the vaccine used for primary vaccination.
  Arms: Pfizer Booster Recommendation

SUMMARY:
While both heterologous (mixing) and homologous (matching) vaccine regimens are now considered standard of care, post-vaccination complications and long-term effects of the different vaccination regimens have not been thoroughly studied. There is a pressing need to investigate the longitudinal effects of the mixing and matching vaccine-booster approaches. This study proposes to utilize the existing digital infrastructure of the COVID-19 Citizen Science (CCS) study on the Eureka Research Platform to perform a systematic and prospective randomized trial comparing mixing versus matching approaches. Eligible CCS participants will have the opportunity to be randomly assigned to a recommendation of receiving either the Pfizer or Moderna booster vaccine. Long-term effects will be monitored through the participants' completion of their regular weekly CCS follow-up surveys on symptoms and infection. This randomized trial aims to mitigate the effect of confounding variables and provide more conclusive evidence on each regiment to guide booster recommendations.

DETAILED DESCRIPTION:
The FDA recently approved the use of COVID-19 booster vaccines for both homologous and heterologous vaccine booster regimens, with both regimens considered standard of care. However, there is incomplete research on the long-term effects and immunity offered by each approach. In fact, the FDA has not offered guidance on whether or not to mix or match vaccines because as of yet, there is no evidence indicating that one strategy should be recommended over the other. Studies have shown that vaccine efficacy declines over time, and the Delta and Omicron variants continue to cause breakthrough cases. Additionally, millions of Americans are now becoming eligible for a booster. These factors present both a pressing need and a unique opportunity to investigate the longitudinal effects of the mixing and matching vaccine-booster approaches.

This study proposes to fill this critical gap through a systematic and prospective randomized trial utilizing the existing digital infrastructure of the COVID-19 Citizen Science (CCS) study on the Eureka Research Platform. Eligible CCS participants will have the opportunity to be randomly assigned to be encouraged to receive either the BNT162b2 (Pfizer) or mRNA-1273 (Moderna) booster vaccine and will continue to complete their weekly CCS follow up surveys on symptoms and infection. Thus, this study will allow for longitudinal follow up of participants receiving homologous and heterologous vaccine booster regimens. By randomizing participants and analyzing a larger cohort, this study aims to mitigate the effect of confounding variables and provide more conclusive evidence to guide booster recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled in the COVID19 Citizen Science (CCS) study. The CCS study is a remote, longitudinal, observational registry hosted on the Eureka Research Platform that administers weekly questionnaires to participants regarding COVID-19 symptoms and exposures. CCS is currently open to enrollment for adults aged 18 and older who have a smartphone device to participate on the mobile app, or an email address to participate on the web portal.
* Must have received either 2 doses of mRNA vaccine such as Moderna and Pfizer, or 1 dose of Johnson and Johnson

Exclusion Criteria:

* Already received a COVID19 booster
* Are not planning on receiving a COVID19 booster in the next 3 months
* Do not have equal access to both the Pfizer and Moderna boosters
* Have a medical reason to receive either the Pfizer or Moderna booster
* Have a medical reason to not receive any booster (e.g h/o allergic reaction to an mRNA vaccine or myocarditis or pericarditis after an mRNA vaccine)
* Are unwilling to be randomized
* Are unable to commit to filling out the CCS weekly surveys consistently (to the best of their ability)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Post-Vaccine Differences in Types of Symptoms between Pfizer and Moderna | 1 year
  The study will assess differences in types of symptoms participants experience post-vaccination between the randomization groups (Pfizer vs. Moderna). The types of symptoms will be assessed through a questionnaire post-vaccination asking participants if they have any of the following symptoms: fever, chills, fatigue, sore/scratchy throat, muscle pain, joint pain, headache, other pain, rash, allergic reaction/anaphylaxis.
Post-Vaccine Differences in Severity of Symptoms between Pfizer and Moderna | 1 year
  The study will assess differences in severity participants experience post-vaccination between the randomization groups (Pfizer vs. Moderna). The severity for each symptom will be assessed through a post-vaccination questionnaire asking participants how many days the participant experienced their symptoms, and how severe their symptoms were on a scale of 1 to 5 (1 being mild, 5 being very severe).
Post-Vaccine Differences in Types of Symptoms between Homologous vs Heterologous Regiments | 1 year
  The study will assess differences in types of symptoms participants experience post-vaccination between people who receive the same type of booster vaccine as their initial series (homologous) and people who receive a different type of booster vaccine than their initial series (heterologous) regiments. The types of symptoms will be assessed through a questionnaire post-vaccination asking participants if they have any of the following symptoms: fever, chills, fatigue, sore/scratchy throat, muscle pain, joint pain, headache, other pain, rash, allergic reaction/anaphylaxis.
Post-Vaccine Differences in Severity of Symptoms between Homologous vs Heterologous Regiments | 1 year
  The study will assess differences in severity of symptoms participants experience post-vaccination between people who receive the same type of booster vaccine as their initial series (homologous) and people who receive a different type of booster vaccine than their initial series (heterologous) regiments. The severity of each symptom will be assessed through a post-vaccination questionnaire asking participants how many days the participant experienced their symptoms, and how severe their symptoms were on a scale of 1 to 5 (1 being mild, 5 being very severe).

SECONDARY OUTCOMES:
COVID-19 Infection Rates between Pfizer and Moderna | 1 year
  The study will compare COVID-19 infection rates among those who receive the Moderna booster vs. the Pfizer booster
COVID-19 Infection Rates between Homologous vs Heterologous Regiments | 1 year
  The study will compare COVID-19 infection rates among those with homologous vs. heterologous vaccine regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Marcus, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Parnassus, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT05268185/ICF_000.pdf